CLINICAL TRIAL: NCT06934265
Title: Phonation Resistance Training Exercises (PhoRTE®) Delivered In-person and Via Telehealth: A Noninferiority Randomized Clinical Trial
Brief Title: PhoRTE® Therapy Efficacy: In-Person Versus Telehealth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Aaron Rothbart, PhD, Clinical Assistant Professor of Otolaryngology - Head and Neck Surgery (Clinician Educator), University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APP-24-06117
Record Dates: First submitted 2025-03-11; First posted 2025-04-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Atrophy of Vocal Cord; Presbyphonia; Dysphonia; Glottic Insufficiency; Voice Change; Voice Disorder; Adults; Aging; Speech Therapy; Voice Alteration
Keywords: Vocal fold atrophy; voice therapy; presbyphonia; aging voice; voice rehabilitation; speech pathology; Intervention; voice; aging
MeSH Terms: conditions — Dysphonia; Voice Disorders; Communication Disorders

STUDY DESIGN:
Intervention Model Description: Each group will get the same intervention; however, delivery method will differ (in-person vs telehealth-delivered)
Who Masked: Investigator
Masking Description: CAPE-V audio sample listeners will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PhoRTE - IP (Active Comparator): PhoRTE® voice therapy will be administered to this treatment arm in-person (IP)(traditional therapy).
  Interventions: Behavioral: exuberant voice therapy
- PhoRTE - TH (Experimental): Study participants who will be receiving intervention via telehealth. Intervention administered will be PhoRTE® voice therapy.
  Interventions: Behavioral: exuberant voice therapy

INTERVENTIONS:
Behavioral: exuberant voice therapy — exuberant voice therapy validated for patients with age-related voice changes (i.e., vocal fold atrophy, presbyphonia)
  Other Names: Phonation Resistance Training Exercises (PhoRTE®)

SUMMARY:
This study compares how well voice therapy works when delivered in-person versus through telehealth for older adults with age-related voice problems. Researchers are testing whether Phonation Resistance Training Exercises (PhoRTE®) can be just as effective when delivered remotely as when done face-to-face, which could make treatment more accessible and affordable for seniors.

The two primary hypotheses are:

1. Does voice therapy (called PhoRTE®) work as well through video calls as it does face-to-face?
2. Can online therapy be a more accessible way for older adults to get help for their voice problems?

Adults aged 55 or older with voice changes and an applicable diagnosis will be randomly assigned to receive either in-person or telehealth therapy, consisting of four 45-minute sessions. After treatment, researchers will measure improvements through:

* Changes in voice function
* Patient reports about their voice
* Scientific measurements of voice quality
* Patient satisfaction with treatment
* Impact on quality of life

The results will help determine if telehealth can be a good alternative to in-person voice therapy, especially important as telehealth coverage may be changing.

DETAILED DESCRIPTION:
This study employs a prospective, noninferiority cohort design to compare the efficacy of in-person versus telehealth delivery of Phonation Resistance Training Exercises (PhoRTE®) for adults aged 55+ diagnosed with presbyphonia.

Participants will be recruited from the USC Voice Center, a multidisciplinary otolaryngology clinic with four outpatient locations in Southern California. Eligible participants must have a primary diagnosis of presbyphonia, age-related voice change, and/or vocal fold atrophy.

The study will use stratified block randomization with a 1:1 allocation ratio to ensure equitable distribution of severity across both treatment groups (in-person and telehealth). Electronic randomization algorithms will be implemented to mitigate selection bias.

Treatment Protocol:

* Both groups will complete four 45-minute sessions of voice therapy
* Sessions will be conducted at weekly or biweekly intervals
* PhoRTE® therapeutic intervention involves exuberant vocalization techniques utilizing high-intensity phonation with expanded oral aperture configuration ("megaphone mouth shape") to optimize phonatory efficiency and augment vocal intensity without inducing vocal strain/hyperfunction

Assessment Measures:

1. Validated patient-reported outcomes:

   1. Voice Handicap Index-10 (VHI-10) for quantification of perceived voice-related quality of life impairment
   2. Aging Voice Index (AVI) for quantification of perceived voice-related quality of life impairment for aging populations
   3. OMNI-Vocal Effort Scale for perceived assessment of effort with voicing
   4. Voice Problem Impact Scales (VPIS) for multidimensional evaluation of voice-related quality of life
2. Expert clinical auditory/perceptual measures:

   Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) for voice quality and severity Note: Blinded independent evaluation by voice & upper airways-specialized (VUAD) speech-language pathologists (minimum 5 years specialization in voice disorders with ≥80% voice disorder caseload) analysis of recorded voice samples
3. Instrumental acoustic/aerodynamic measures:

   1. Acoustic measures: cepstral peak prominence (CPP), CPP standard deviation (CPP SD), fundamental frequency (fo), and vocal intensity/loudness (dB SPL) in sustained vowels and connected speech - Aerodynamic measures: subglottal pressure (Psub), phonation threshold pressure (PTP), and mean airflow during voicing with corresponding duration and number of replenishing breaths during sustained vowels and connected speech

Data Collection Timeline:

* Baseline measures will be obtained at the initial interprofessional evaluation
* Post-intervention evaluations will occur one week after the terminal therapeutic session
* All measurement parameters will be repeated at both timepoints to assess treatment effects

Sample Size:

The target enrollment is 13-15 participants per treatment group (26-30 participants total), which aligns with previous research on PhoRTE® therapy for presbyphonia.

This protocol follows the tripartite model of evidence-based practice and therefore contains multiple primary outcomes through integration of patient-reported measures, clinical expertise, and instrumental assessment to comprehensively evaluate treatment efficacy across delivery modalities.

ELIGIBILITY:
Inclusion Criteria:

* Adults 55+ with a primary diagnosis of presbyphonia, age-related voice changes, and/or vocal fold atrophy with or without localized loss of lamina propria (e.g. vocal fold scar)
* Telehealth-capable device (e.g., tablet, computer) with microphone, speaker, camera, high-speed internet
* Ability to attend four telehealth or in-person sessions for four consecutive sessions
* Ability to attend two in-person evaluation sessions (pre- and post-treatment)

Exclusion Criteria:

* Presence of localized masses, lesions, or vocal fold motion impairments identified during videostroboscopy at initial evaluation
* Progressive neurologic conditions, e.g. Parkinson's disease (PD), Amyotrophic lateral sclerosis (ALS), Progressive supranuclear palsy (PSP), etc.
* Previous attendance to exuberant voice therapy (e.g., PhoRTE, Lee Silverman Voice Treatment)
* Untreated hearing loss
* Non-English speakers

Min Age: 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-07-25 (Estimated); Study Completion 2026-10-25 (Estimated)

PRIMARY OUTCOMES:
Voice Handicap Index-10 | up to 16 weeks
  5 point likert scale to assess voice-related quality of life impairment, where 0 = never, 1 = almost never, 2 = sometimes, 3 = almost always, 4 = always. 10 questions in total. Higher score indicates a greater voice handicap. Score of >11 is considered abnormal. Measure will be collected at initial evaluation (baseline) and again following intervention (final evaluation).
Aging Voice Index | up to 16 weeks
  AVI Score at Baseline and re-evaluation. The Aging Voice Index (AVI) is a validated instrument that measures quality of life in older adults with voice disorders. A higher score indicates worse quality of life. Scores range from 0 to 92.
Voice Problem Impact Scales | up to 16 weeks
  A validated self assessment questionnaire in which the participant self-rates impact of voice on four domains of life on 1-7 likert scales (1. work/daily activities, 2. social life, 3. home life, 4. life overall.) Numbers are presented in equally appearing intervals with end anchors where 1=not at all affected and 7=profoundly. A higher score indicates higher degree of impact.
  Measure will be collected at initial evaluation (baseline) and again following intervention (final evaluation).
Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) | up to 16 weeks
  A validated auditory/perceptual voice quality and severity assessment tool to be used pre- and post-intervention. Blinded independent expert clinicians, identified as SLPs who have 5+ years of experience in the assessment and treatment of patients with voice disorders and who currently maintain a caseload of at least 80% voice patients, will assess recorded voice samples to describe participant voice quality and severity using the CAPE-V.
  Measure will be collected at initial evaluation (baseline) and again following intervention (final evaluation).
OMNI Vocal Effort Scale | up to 16 weeks
  Visual analog scale for patient-perceived vocal effort on a 0-10 scale where 0=extremely easy and 10=extremely hard. Patient is asked for perception of current voice effort during assessment and highest effort level experienced.
Acoustic Assessment: voicing intensity | up to 16 weeks
  Acoustic measure in sustained voicing via mean intensity (in dB SPL) and its standard deviation across a. standardized vowel /a/, b. standardized reading passage (Rainbow passage), and c. running, conversational speech.
  Measure will be collected at initial evaluation (baseline) and again following intervention (final evaluation).
Acoustic Assessment: Cepstral Peak Prominence | up to 16 weeks
  Acoustic measure in sustained voicing using Cepstral Peak Prominence and its standard deviation while reading a standardized passage (Rainbow passage).
  Measure will be collected at initial evaluation (baseline) and again following intervention (final evaluation).
Aerodynamic Measurement: phonatory airflow during speech | up to 16 weeks
  Airflow during voicing will be measured at baseline and again at final evaluation using the Phonatory Aerodynamic System Model 6600 (PAS; PENTAX Medical). Assessment includes flow during voicing across a. sustained vowel /a/ and running speech (first four sentences of standardized Rainbow Passage).
  The PAS reports airflow during voicing using a pneumotach with integrated facemask and external microphone. During voicing, pressure transducers on either side of the terminal collects and converts the air flow across time to determine airflow rate. The microphone captures the acoustic signal according to terminal-specific standardized calibration. Subjects maintain upright seated posture with the face mask firmly pressed to their face, ensuring an airtight seal over oral and nasal cavities during this task.
Aerodynamic Measurement: subglottal pressure | up to 16 weeks
  Subglottal pressure (Psub) will be measured at initial evaluation (baseline) and again at the conclusion of therapeutic intervention (final evaluation) using the Phonatory Aerodynamic System Model 6600 (PAS; PENTAX Medical). Assessment utilizes the valid labial interruption task via /pipipi/ syllable production task.
  The PAS collects intraoral pressure, which is a validated, non-invasive approximate to subglottal pressure. The participant thens produce the sequence at a comfortable pitch and loudness. Analysis then extracts the subglottal pressure by measuring airflow and intraoral pressure during speech.
Aerodynamic Measurement: phonation threshold pressure | up to 16 weeks
  Phonation threshold pressure (PTP) will be measured at initial evaluation (baseline) and again at the conclusion of therapeutic intervention (final evaluation) using the Phonatory Aerodynamic System Model 6600 (PAS; PENTAX Medical). Assessment utilizes the valid labial interruption task via /pipipi/ syllable production. PTP is the minimum subglottal pressure required to initiate and sustain vocal fold oscillation.
  The PAS collects intraoral pressure, which is a validated, non-invasive approximate to subglottal pressure. The participant thens produces the sequence at their softest vocal intensity. Analysis extracts the PTP by measuring the relationship between airflow and intraoral pressure at softest possible voicing.
Aerodynamic Measurement: number of breaths | up to 16 weeks
  mean number of breaths across a standardized reading passage (The Rainbow Passage) collected at baseline (initial evaluation) and once again after intervention (final evaluation).
duration across standardized reading passage | up to 16 weeks
  mean duration (in seconds) to complete the reading of a standard passage (The Rainbow Passage).

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Rothbart, PhD, Principal Investigator — University of Southern California
Locations (4):
- United States (4):
  - USC Voice Center, Arcadia, California
  - USC Voice Center, Beverly Hills, California
  - USC Voice Center, Glendale, California
  - USC Voice Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No
The number of resources and collaboration to collect and analyze the data is not feasible for the current research question and current available time and funding.

REFERENCES:
- [Background] Shoffel-Havakuk H, Marks KL, Morton M, Johns MM 3rd, Hapner ER. Validation of the OMNI vocal effort scale in the treatment of adductor spasmodic dysphonia. Laryngoscope. 2019 Feb;129(2):448-453. doi: 10.1002/lary.27430. Epub 2018 Oct 12. PMID 30315575
- [Background] Galluzzi F, Garavello W. The aging voice: a systematic review of presbyphonia. Eur Geriatr Med. 2018 Oct;9(5):559-570. doi: 10.1007/s41999-018-0095-6. Epub 2018 Sep 3. PMID 34654233
- [Background] Desjardins M, Halstead L, Simpson A, Flume P, Bonilha HS. Respiratory Muscle Strength Training to Improve Vocal Function in Patients with Presbyphonia. J Voice. 2022 May;36(3):344-360. doi: 10.1016/j.jvoice.2020.06.006. Epub 2020 Jul 14. PMID 32680804
- [Background] Lindstrom E, Ohlund Wistbacka G, Lotvall A, Rydell R, Lyberg Ahlander V. How older adults relate to their own voices: a qualitative study of subjective experiences of the aging voice. Logoped Phoniatr Vocol. 2023 Dec;48(4):163-171. doi: 10.1080/14015439.2022.2056243. Epub 2022 Apr 21. PMID 35446741
- [Background] Ziegler A, Verdolini Abbott K, Johns M, Klein A, Hapner ER. Preliminary data on two voice therapy interventions in the treatment of presbyphonia. Laryngoscope. 2014 Aug;124(8):1869-76. doi: 10.1002/lary.24548. Epub 2014 Jan 29. PMID 24375313
- [Background] Guglani I, Sanskriti S, Joshi SH, Anjankar A. Speech-Language Therapy Through Telepractice During COVID-19 and Its Way Forward: A Scoping Review. Cureus. 2023 Sep 6;15(9):e44808. doi: 10.7759/cureus.44808. eCollection 2023 Sep. PMID 37809138
- [Background] Griffin M, Bentley J, Shanks J, Wood C. The effectiveness of Lee Silverman Voice Treatment therapy issued interactively through an iPad device: A non-inferiority study. J Telemed Telecare. 2018 Apr;24(3):209-215. doi: 10.1177/1357633X17691865. Epub 2017 Feb 1. PMID 28147896
- [Background] Theodoros DG, Hill AJ, Russell TG. Clinical and Quality of Life Outcomes of Speech Treatment for Parkinson's Disease Delivered to the Home Via Telerehabilitation: A Noninferiority Randomized Controlled Trial. Am J Speech Lang Pathol. 2016 May 1;25(2):214-32. doi: 10.1044/2015_AJSLP-15-0005. PMID 27145396
- [Background] Titze IR, Palaparthi A, Cox K, Stark A, Maxfield L, Manternach B. Vocalization with semi-occluded airways is favorable for optimizing sound production. PLoS Comput Biol. 2021 Mar 29;17(3):e1008744. doi: 10.1371/journal.pcbi.1008744. eCollection 2021 Mar. PMID 33780433
- [Background] Belsky MA, Shelly S, Rothenberger SD, Ziegler A, Hoffman B, Hapner ER, Gartner-Schmidt JL, Gillespie AI. Phonation Resistance Training Exercises (PhoRTE) With and Without Expiratory Muscle Strength Training (EMST) For Patients With Presbyphonia: A Noninferiority Randomized Clinical Trial. J Voice. 2023 May;37(3):398-409. doi: 10.1016/j.jvoice.2021.02.015. Epub 2021 Mar 16. PMID 33741235
- [Background] Kempster GB, Gerratt BR, Verdolini Abbott K, Barkmeier-Kraemer J, Hillman RE. Consensus auditory-perceptual evaluation of voice: development of a standardized clinical protocol. Am J Speech Lang Pathol. 2009 May;18(2):124-32. doi: 10.1044/1058-0360(2008/08-0017). Epub 2008 Oct 16. PMID 18930908
- [Background] Castro ME, Sund LT, Hoffman MR, Hapner ER. The Voice Problem Impact Scales (VPIS). J Voice. 2024 May;38(3):666-673. doi: 10.1016/j.jvoice.2021.11.011. Epub 2021 Dec 20. PMID 34933795
- [Background] Rosen CA, Lee AS, Osborne J, Zullo T, Murry T. Development and validation of the voice handicap index-10. Laryngoscope. 2004 Sep;114(9):1549-56. doi: 10.1097/00005537-200409000-00009. PMID 15475780
- See also: Intervention approach website — https://www.phorte.org/